CLINICAL TRIAL: NCT00107536
Title: A Phase II Study of Efficacy and Tolerability of GW572016 in Patients With Advanced Hepatocellular and Biliary Carcinomas
Brief Title: Lapatinib Ditosylate in Treating Patients With Unresectable Liver or Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01464; OSU 0447; N01CM62207 (NIH); N01CM62201 (NIH); CDR0000420830 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-03

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Arm I (Experimental): Patients receive oral lapatinib ditosylate once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This phase II trial is studying how well lapatinib ditosylate works in treating patients with unresectable liver or biliary tract cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate (complete response [CR] + partial response [PR]) as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria in each group of patients.

SECONDARY OBJECTIVES:

I. To evaluate the progression free survival at 6 months. II. To evaluate the toxicity profile of this treatment in each group of patients.

III. To evaluate median overall survival, 6 and 12 months survival rates. IV. To assess target-epidermal growth factor receptor (EGFR)/EGFR-P protein expression and the genes that regulate the cell cycle and apoptosis, which are either downstream of or cross-talk with the EGFR signaling pathway, to explore their association with clinical outcome.

V. To measure expression profile and mutations of genes critical for EGFR and (v-erb-b2 erythroblastic leukemia viral oncogene homolog 2 (ERBB2 signaling pathways with particular relevance to GW572016, and to explore new gene-drug relationships as relating to hepatocellular and biliary carcinomas.

OUTLINE: This is a multicenter study.

Patients receive oral lapatinib ditosylate once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following:

  * Hepatocellular carcinoma (hepatoma)

    * Child-Pugh classification score ≤ 7
  * Biliary tract carcinoma
* Surgically unresectable disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Fresh tissue or paraffin embedded tissue from tumor blocks available
* No ampulla of Vater tumors
* No known brain metastases
* Performance status - ECOG 0-1
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Albumin ≥ 2.5 mg/dL
* INR ≤ 1.5 (for patients not receiving an anticoagulant)
* Live metastases or stable chronic liver disease allowed
* No current active hepatic or biliary disease except for Gilbert's syndrome or asymptomatic gallstone
* Creatinine ≤ 2 mg/dL
* Ejection fraction normal by echocardiogram or MUGA
* No unstable angina pectoris
* No cardiac arrhythmia
* Able to swallow and retain oral medication
* No gastrointestinal (GI) tract disease resulting in an inability to take oral medication
* No malabsorption syndrome
* No requirement for IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant traumatic injury within the past 3 weeks
* No active or ongoing infection
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to lapatinib
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* More than 4 weeks since prior biologic therapy
* More than 4 weeks since prior immunotherapy
* See Radiotherapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior cumulative doxorubicin dose > 450 mg/m^2
* At least 14 days since prior and no concurrent glucocorticoids (e.g., dexamethasone or equivalent [dose > 1.5 mg/day])
* More than 4 weeks since prior radiotherapy
* More than 12 weeks since prior radiotherapy with or without a fluoropyrimidine as a radiosensitizer (for patients with biliary carcinoma only)
* No prior surgical procedure affecting absorption
* More than 3 weeks since prior major surgery
* Recovered from all prior therapy
* No more than 1 prior systemic anticancer therapy, including chemoembolization
* No prior epidermal growth factor receptor-targeting therapy
* More than 6 weeks since prior cryotherapy, radiofrequency ablation, ethanol injection, transarterial chemoembolization, or photodynamic therapy AND meets both of the following criteria:

  * Indicator lesion is outside the area of prior treatment OR there is clear evidence of disease progression associated with the sole indicator lesion
  * Edges of indicator lesion are clearly distinct by CT scan
* At least 7 days since prior and no concurrent H2 inhibitors or proton pump inhibitors

  * Concurrent antacids allowed provided they are administered > 1 hour before and > 1 hour after study drug administration
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following:

  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Delaviridine
  * Ritonavir
  * Indinavir
  * Saquinavir
  * Nelfinavir
  * Amprenavir
  * Lopinavir
  * Itraconazole
  * Ketoconazole
  * Voriconazole
  * Fluconazole (doses ≤ 150 mg/day are allowed)
  * Nefazodone
  * Fluvoxamine
  * Verapamil
  * Diltiazem
  * Cimetidine
  * Aprepitant
  * Grapefruit and grapefruit juice
  * Bitter orange
* At least 6 months since prior and no concurrent amiodarone
* At least 14 days since prior and no concurrent CYP3A4 inducers, including any of the following:

  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Oxcarbazepine
  * Efavirenz
  * Nevirapine
  * Rifampin
  * Rifabutin
  * Rifapentine
  * Roxithromycin
  * Telithromycin
  * Hypericum perforatum (St. John's wort)
  * Modafinil
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* Concurrent oral anticoagulants (e.g., coumadin or warfarin) allowed provided there is increased vigilance in monitoring INR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Bekaii-Saab, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Peck J, Wei L, Zalupski M, O'Neil B, Villalona Calero M, Bekaii-Saab T. HER2/neu may not be an interesting target in biliary cancers: results of an early phase II study with lapatinib. Oncology. 2012;82(3):175-9. doi: 10.1159/000336488. Epub 2012 Mar 15. PMID 22433475
- [Result] Bekaii-Saab T, Markowitz J, Prescott N, Sadee W, Heerema N, Wei L, Dai Z, Papp A, Campbell A, Culler K, Balint C, O'Neil B, Lee RM, Zalupski M, Dancey J, Chen H, Grever M, Eng C, Villalona-Calero M. A multi-institutional phase II study of the efficacy and tolerability of lapatinib in patients with advanced hepatocellular carcinomas. Clin Cancer Res. 2009 Sep 15;15(18):5895-901. doi: 10.1158/1078-0432.CCR-09-0465. Epub 2009 Sep 8. PMID 19737952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between the dates of March 3, 2006-May 14, 2007.
Groups:
- Lapatinib: Patients receive oral lapatinib ditosylate once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  lapatinib ditosylate
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Lapatinib
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients receive oral lapatinib ditosylate once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  lapatinib ditosylate
  laboratory biomarker analysis: Correlative studies
Arm/Group | Arm I
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 58 [29 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 26
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG Performance status 0 is defined as fully active, able to carry on all pre-disease performance without restriction
  ECOG Performance status 1 is defined as restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  participants
    Performance status 0 | 12
    Performance status 1 | 14
Sites of metastasis [Number; unit: participants]
  Lymph nodes | 8
  Lungs | 8
  Spine | 1
  Bone | 1
  Adrenal gland | 1
  Peritoneal mets | 1
  Hepatic mets | 1
  Chest wall | 1
  Not available | 4
Prior treatments [Number; unit: participants]
  X-ray treatment | 3
  Chemo-embolization | 2
  Surgery | 16
  Chemotherapy | 3
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Demonstrating Objective Response (PR+CR) as Defined by RECIST
Description: PR (Partial Response) definded as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. CR (Complete Response) is defined as the disappearance of all target lesions.
Time Frame: Up to 3 years
Population: Only 25 patients were evaluable for response (1 patient passed away before staging).
Measure: Number; unit: patients
Arm/Group | Arm I
Number analyzed (Participants) | 25
patients | 0

2. Secondary Outcome: Progression-free Survival
Time Frame: up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 26
months | 1.9 [1.8 to 3.6]

3. Secondary Outcome: Toxicity Profile Assessed Using NCI CTCAE Version 3.0
Description: Percentage of patients with Adverse events accordng to NCI CTCAE version 3.0
Time Frame: Up to 3 years
Population: All 26 patients were evaluable for toxicity analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Arm I
Number analyzed (Participants) | 26
percentage of patients
  Diarrhea | 73
  Nausea | 54
  Rash | 50

4. Secondary Outcome: Median Overall Survival
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 26
months | 12.6 [7.8 to 22.4]

5. Secondary Outcome: Overall Survival
Time Frame: up to 12.6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 26
months | 12.6 [7.8 to 22.4]

6. Secondary Outcome: Target-EGFR/EGFR-P Protein Expression
Description: EGFR (exons 18-21)
Time Frame: Up to 3 years
Measure: Number; unit: patients with somatic mutations
Arm/Group | Arm I
Number analyzed (Participants) | 26
patients with somatic mutations | 0

7. Secondary Outcome: Expression Profile and Mutations of Genes Critical for EGFR and ERBB2 Signaling Pathways
Time Frame: Up to 3 years
Measure: Number; unit: patients with mutations
Arm/Group | Arm I
Number analyzed (Participants) | 24
patients with mutations | 0

ADVERSE EVENTS:
Time Frame: Week 1 through end of study evaluation
Description: The NCI Common Terminology Criteria for Adverse Events v3.0 was utilized for Adverse Event (AE) reporting.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 26/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=26)
Diarrhea (Gastrointestinal disorders) | 19 (19) — Grade 1, 2, 3
Nausea (Gastrointestinal disorders) | 14 (14) — Grade 1, 2, 3
Fatigue (General disorders) | 11 (11) — Grade 1, 2, 3
Vomiting (Gastrointestinal disorders) | 7 (7) — Grade 1, 2, 3
Alkaline phosphatase (Investigations) | 5 (5) — Grade 1, 2, 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5 (5) — Grade 1, 2, 3
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 4 (4) — Grade 1, 2, 3
Hemoglobin (Blood and lymphatic system disorders) | 4 (4) — Grade 1, 2, 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (3) — Grade 1, 2, 3
Leukocytes (total WBC) (Investigations) | 2 (2) — Grade 1, 2, 3
Anorexia (Metabolism and nutrition disorders) | 3 (3) — Grade 1, 2, 3
Creatinine (Investigations) | 2 (2) — Grade 1, 2, 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2) — Grade 1, 2, 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2) — Grade 1, 2, 3
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2 (2) — Grade 1, 2, 3
Rash (Skin and subcutaneous tissue disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less